CLINICAL TRIAL: NCT02081118
Title: A Phase II, 16-week, Double-blind, Placebo-controlled, Parallel-group, Randomised, Multicentre Trial to Assess Effect on Glycaemic Control of Three Doses of HM11260C in Subjects With Inadequately Controlled Type 2 Diabetes Receiving a Stable Dose of Metformin
Brief Title: Glycaemic Control of Monthly LAPS-Exendin Versus Placebo in Subjects of Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-EXC-204
Record Dates: First submitted 2014-02-24; First posted 2014-03-07 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- HM11260C (8 mg) (Experimental): Monthly administration of 8 mg of HMC11260C by subcutaneous injection for 16 weeks
  Interventions: Drug: HM11260C
- HM11260C (12 mg) (Experimental): Monthly administration of 12 mg of HMC11260C by subcutaneous injection for 16 weeks
  Interventions: Drug: HM11260C
- HM11260C (16 mg) (Experimental): Monthly administration of 16 mg of HMC11260C by subcutaneous injection for 16 weeks
  Interventions: Drug: HM11260C
- Placebo (Placebo Comparator): Monthly administration of placebo by subcutaneous injection for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HM11260C — HM11260C is a novel long-acting form of CA Exendin-4 (an Exendin-4 analogue)
  Other Names: LAPS-Exendin-4
  Arms: HM11260C (12 mg); HM11260C (16 mg); HM11260C (8 mg)
Drug: Placebo — Placebo for HM11260C
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the optimal dose or doses of HM11260C, when administered once a month under the skin, to improve the control of blood sugar levels in patients with early-stage type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study : 18 years to 74 years
* Genders eligible for study : Male and Female
* Diagnosed with T2DM
* Taking a stable dose of metformin monotherapy
* HbA1c levels of between ≥ 7.0% and ≤ 10.0%
* Females of childbearing potential who are not pregnant and agree to use a reliable method of birth control
* Written informed consent must be obtained

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Diagnosis of type 1 diabetes mellitus
* Uncontrolled diabetes defined as a FPG level of > 240 mg/dL at screening
* A significant change in body weight in the 3 months before screening
* Any history of GI intolerance
* Personal or family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC
* Known history of acute or chronic pancreatitis
* A history of alcohol or drug abuse or drug addiction

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in baseline in glycosylated haemoglobin (HbA1c) at 16 weeks | Up to day 155

SECONDARY OUTCOMES:
Fasting plasma glucose levels (FPG) | Up to day 155
7-point glucose profile | Up to day 155
Serum lipid profile | Up to day 155
Body weight | Up to day 155
Fasting insulin | Up to day 155
C-peptide | Up to day 155
Glucagon | Up to day 155
Glycated albumin | Up to day 155

OTHER OUTCOMES:
Number of Participants with Adverse Events by HM11260C | Up to day 155
Number of Participants with Immunogenicity by HM11260C | Up to day 155

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi pharmaceutical, Miami, Florida, United States